CLINICAL TRIAL: NCT04812639
Title: Buccal Infiltration Technique in Comparison to the Inferior Alveolar Nerve Block Technique for Anesthetizing Mandibular Primary Molars During Pulpal Treatment
Brief Title: Buccal Infiltration Technique Compared to Inferior Alveolar Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Sherif Ahmed Abo El Abbas, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BI vs IANB
Record Dates: First submitted 2021-03-14; First posted 2021-03-23 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Local Anesthetic Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: not showing the anesthetic procedure in the video tape
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buccal infiltartion technique (Experimental): local anesthetic technique
  Interventions: Other: Inferior alveolar nerve block technique
- Inferior alveolar nerve block technique (Active Comparator): local anesthetic technique
  Interventions: Other: Buccal infiltration technique

INTERVENTIONS:
Other: Buccal infiltration technique — a technique for injecting local anesthetic solution in the buccal mucobuccal fold between the roots of the targeted tooth
  Arms: Inferior alveolar nerve block technique
Other: Inferior alveolar nerve block technique — a technique for injecting local anesthetic solution to anesthetize the inferior alveolar nerve
  Arms: buccal infiltartion technique

SUMMARY:
This study was conducted to compare the efficacy of the buccal infiltration technique with inferior alveolar nerve block technique for alleviation of intraoperative pain during pulpal treatment of second mandibular primary molars using 4% Articaine 1:100000.

The study started with 22 cooperative medically free patients aging 7 to 8 years old seeking treatment for bilateral deep carious mandibular second primary molars with no previous history of irreversible pulpitis, swelling, sinus tract or tooth mobility.

Randomization was achieved when each candidate was instructed to pick an opaque and sealed envelope from two separate black and opaque boxes. First box contained two envelopes to identify the side on which the operator will perform the treatment. While the second box contained another two envelopes describing which anesthetic technique will be implemented with the previously chosen side.

After clinical and radiographic examination, the patient received the pulpal treatment under the identified side and injecting technique. Videotaping of the pulpal treatment procedure was initiated after numbness was experienced by the child.

A blind assessor was assigned to review the videos and fill in the SEM pain scale to identify the pain and level of discomfort experienced by the child during the pulpal treatment.

DETAILED DESCRIPTION:
This study was a split mouth randomized controlled trial enrolling 22 patients from the diagnostic center in the Pediatric Dentistry and Dental Public Health Department Faculty of Dentistry, Cairo University. All participants met the following inclusion criteria:

1. Cooperative children (rating four or three based on Frankl behavior scale) aging from seven to eight years.
2. Medically free child categorized as ASA I or ASA II according to the American Society of anesthesiologist.
3. Restorable bilateral deep carious lower primary second molars as shown in figure (1).
4. Normal radiographic findings.

Preoperative periapical x-rays were done on the targeted molars to confirm their adherence to the eligibility criteria and to confirm their restorability.

Each participant was asked to pick an opaque and sealed envelope from two separate black and opaque boxes to randomly choose the operated technique and side on the first operating visit. By default the other technique will be implemented on the other side on the upcoming visit.

Proper psychological management and desensitization procedures were undertaken to prepare the patient for the treatment. Certain phrases were used to prepare the child for applying topical anesthetic gel and injecting the anesthetic agent in any given technique like "The magic water will be used to put the tooth to sleep".

The protocols followed for inferior alveolar nerve block and buccal infiltration techniques were according to Jones and Dean; 2016 and Tudeshchoie et al; 2013.

Caries removal and pulpal treatment were videotaped with both local anesthetic techniques. Caries was removed using a high speed contra with copious cooling and proper suction, complete deroofing and excavation to the coronal pulpal tissues, bleeding from canals was evaluated after the application of a wet cotton for two to four minutes, and then a cotton damped with formocresol was applied for two to four minutes, fixation and brown stumps had to be evident for applying the zinc oxide and eugenol dressing in the pulp chamber.

If any pain was felt during the procedure and the patient raised his/her left hand the procedure was immediately halted. If pulpal exposure was still not evident additional anesthesia was injected through the inferior alveolar nerve block technique since it is the gold standard for anesthetizing mandibular posterior teeth. While if pain was experienced after pulpal exposure few drops of anesthesia was injected intra-pulpally, in both cases and this was considered a failure in the anesthetic technique used.

After application of zinc oxide and eugenol cement, video recording was halted, zinc phosphate cement was then used to seal the coronal part of the tooth and then the tooth was covered with a preformed stainless steel crown.

Videos were then assessed by an assessor who was completely blinded from the technique of injection to fill in a printed (SEM) pain scale sheet for each technique with each participant.

Postoperative instructions were verbally stated to the parent/guardian regarding precautions towards lip biting due to lip numbness. The patient was dismissed, and after at least a week the patient would be recalled to operate on the contralateral side.

In order to ensure complete blindness of the statistician to the results of the local anesthetic techniques, the inferior alveolar nerve block technique (IANB) was designated as Treatment Group I and buccal infiltration technique (BI) was designated as Treatment Group II.

B. Data measurement:

SEM Pain Scale was used to evaluate the intraoperative pain experienced during pulpal treatment of mandibular primary second molars with both local anesthetic techniques using articaine four percent solution.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative children (rating 4 or 3 based on Frankl behavior scale) aging from 7 to 8.
2. Medically free child ASA I or ASA II according to the American Society of anesthesiologist.
3. Restorable bilateral deep carious lower primary second molars.
4. Normal radiographic findings.

Exclusion Criteria:

* 1- Uncooperative child (rating 1 or 2 on the Frankl behavior scale). 2- Signs and symptoms of irreversible pulpitis, spontaneous pain, necrosis or any signs and symptoms of abscess.

  3- Radiographic signs of abscess, bone loss, internal or external root resorption was evident.

  4- Parents or guardians refused participating in the study.

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain during pulpal treatment | up to one month
  Sound Eye Motor SEM Pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Saber H Mohamed, Associate Professor, Study Director — Cairo U
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No